CLINICAL TRIAL: NCT04281225
Title: Mindfulness Intervention and Symptom Variability in Hearing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: With COVID, we are not able to conduct any in-person research at this time
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Ellen Langer, Professor, Harvard University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB19-0222
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Hearing Loss
Keywords: attention to variability; placebo; hearing
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Research Assistants are blind to the conditions of the participants. Participants do not know which condition they have been assigned to either. Only the main investigators (Deb Phillips, Neha Dhawan, Kris Nichols, and Francesco Pagnini) will know which participant is assigned to a particular intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo only condition (Placebo Comparator): Participants in this condition will be told at the time of the initial assessments (T1) that the device they will be testing will improve their hearing. All participants will be instructed to put on the hearing device and listen to an audio twice per day for 6 days. After listening to the 2nd audio of the day, they will be asked if they perceive their hearing to be changed by the device in addition to qualitative descriptions of the audio. This group will allow researchers to investigate the main effect of the placebo hearing aid - without calling participant's attention to variability in their symptoms.
  Interventions: Other: Placebo
- Placebo and ATV condition (Experimental): Participants in this condition at the time of the initial assessments (T1) will be told that the device they will be testing will improve their hearing. They will then be told that in-order to receive the maximum benefit from the hearing device, they should focus on instances in which they can hear better and worse. All participants will be instructed to put on the hearing device and listen to an audio twice per day for 6 days. After listening to the 2nd audio of the day, they will asked 1) if they perceive their hearing to be changed by the device; 2) to note any changes in what they heard in the audio focusing on the story in the ballad; and 3) whether their hearing is possibly impacted by activities and behavior and what they were doing.This condition will enable researchers to test the effects of the interaction between attention to variability and the placebo effect.
  Interventions: Behavioral: Attention to Variability (ATV); Other: Placebo
- ATV only condition (Experimental): Participants in this condition will be told that the device they will be testing is merely a prototype that they are testing for design purposes. However, these participants will also be told that their input while wearing the device will help the team in developing the final device and allow the team to focus on how to best improve hearing. All participants will be instructed to put on the hearing device and listen to an audio twice per day for 6 days. After listening to the 2nd audio of the day, they will be asked 1) to note any changes in what they heard in the audio focusing on the story in the ballad and 2) whether their hearing might possibly be impacted by activities and behavior. They will also be asked 3) about their general health and wellness, as compared to the last time they were contacted by email. This condition will enable researchers to test the main effect of attention to variability, without an explicit placebo effect.
  Interventions: Behavioral: Attention to Variability (ATV)
- Control condition- no ATV or Placebo effect. (No Intervention): Participants in this condition will be told that the device they will be testing is merely a prototype that they are testing for ergonomic purposes. They will listen to the audio and record volume levels at the start and at the end of the audio and provide feedback on the design. They will be told that each day they will listen to a brief audio (ballad of under 3 minutes) and will be asked a few similar questions twice daily for 6 days. After the 2nd audio of the day, they will be asked for feedback on the hearing device design. They will also be asked about their general health and wellness, as compared to the last time they were contacted.This group will allow researchers to test for the effects of having any device at all.

INTERVENTIONS:
Behavioral: Attention to Variability (ATV) — In Attention to Variability we ask the participant to attend to the natural fluctuations in mood and behavior that occur throughout the day, and to notice changes they experience with their hearing loss symptoms; noticing if it is better or worse and to ask why it may be.
  Arms: ATV only condition; Placebo and ATV condition
Other: Placebo — Participants are told that the device they will be testing will improve their hearing, when in fact the device is not a hearing aid but just a metallic earring.
  Arms: Placebo and ATV condition; Placebo only condition

SUMMARY:
The purpose of this study is to investigate the efficacy of mindfulness and placebo treatments on hearing improvement. More specifically, the researchers will be investigating whether the following variables impact the effectiveness of placebo treatment such as: mindfulness, and attention to variability. Extant research has found the effectiveness of psychological treatment in multiple domains, and the researchers look to further investigate this success in the domain of hearing symptom sensations.

DETAILED DESCRIPTION:
The placebo effect, described as "psychological or physiological responses attributed to expectations of an inert substance or procedure, has been demonstrated to have powerful effects in multiple instances (Colloca & Benedetti, 2005). Although research on the placebo effect is prolific, the mechanisms involved can vary based on the context and have been difficult to research with consistent approaches and results (Brown et al., 2013; Holmes et al., 2018). Some researchers have found that the mere perception of a treatment as "new" is enough to elicit a placebo effect, while others have found that the key mechanism may be attention to symptoms - nevertheless, "little evidence exists on the precise mechanisms through which psychological treatments actually work" (Brown et al., 2013; Holmes et al., 2018).

Earlier work suggests the potential for psychological treatments for hearing loss or other forms of hearing disability, including coping techniques (Scott et al, 2009). This study aims to extend the mind-body unity theory as suggested by Dawes et al. (2013) who found in two successive studies that there is a reliable placebo effect in hearing-aid trials. While the objective of these studies was to encourage double-blind methodology (to optimize results), these results suggest that such effects can optimize outcomes and as the audiology field does not typically consider placebo effects. it suggests that hearing improvements can be impacted by (positive) expectations in a "general" sense (not a specific type of hearing aid but simply a "new technology" hearing aid). While this will be of great use clinically in double blind trials, it suggests that the use of a psychological construct, specifically the Langerian attention to variability construct, can function to encourage a placebo effect or a clinical response by encouraging a sense of personal control over the symptoms of the hearing loss. In this study, researchers will look to further investigate one potential mechanism important to the placebo effect - attention to variability.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 80 years of age
* Eyesight with corrective lenses sufficient enough to read and respond to emails
* Owns or has access to and is familiar with using a smartphone and/or desk top/laptop with a cellular data plan and email host
* Able to receive and respond to text messages and emails
* Able to and access to watch, listen to and operate on a phone or computer a video or recording
* English speaking and reading at 8th grade level
* Self-Perceived mild to moderate hearing problem with onset after age 18 (adult onset)

Exclusion Criteria:

* Under age 18 or over age 80
* Unable to read and respond to texts or emails
* No Smartphone or desktop/laptop access
* Hearing loss onset prior to age 18
* Co-morbid conditions such as cancer, diabetes, cardiovascular disease diagnosed and under treatment in the past 6 months
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Hearing Change - subjective preferred volume | 5 minutes daily for 6 days
  Participants will be told to wear the hearing device and listen to a brief audio (ballad of under 3 minutes) twice a day daily for 6 days.The survey will ask them to listen to the audio and record the volume level that they used at the beginning and at the end, and then answer a few questions after. The change in participants subjective preferred volume over the course of the week , compared to T1 at the beginning of the week, will represent hearing change.

SECONDARY OUTCOMES:
Langer Mindfulness Scale,14-Item scale | 5 minutes
  3 subscales, each ranging from 1-7, with 1 being 'Strongly Disagree' and 7 being 'Strongly Agree'. Subscales are 'Flexibility'; 'Novelty Seeking'; and 'Novelty Producing'.Ratings on these items are then added together to create a score for each subscale and an overall mindfulness score. Higher scores indicate greater mindfulness, and can range from 14 to 98.
Perceived Stress Scale (PSS) | 5 minutes
  This 10 item scale asks questions about one's feelings and thoughts during the past month. In each question, individuals are asked how often they felt or thought a certain way on a scale from 0 (Never) to 4 (Very Often). Scores can range from 0 to 40, with a greater values is indicating greater perceived stress.
  Scoring: Each item is rated on a 5-point scale ranging from (0) never to (4) almost always
Hearing Handicap Inventory for Elderly- Screening (HHIE-S) | 5 minutes
  For participants over the age of 65. The Hearing Handicap Inventory for the Elderly Screening Version (HHIE-S) is a 10-item questionnaire that assesses how an individual perceives the social and emotional effects of hearing loss. The higher the HHIE-S score, the greater the handicapping effect of a hearing impairment. Possible scores range from 0 (no handicap) to 40 (maximum handicap).
Hearing Handicap Inventory for Adults- Screening (HHIA-S) | 5 minutes
  Similar to the HHIE-S above but for adult participants under the age of 65. The higher the HHIA- S score, the greater the handicapping effect of a hearing impairment. Possible scores range from 0 (no handicap) to 40 (maximum handicap).

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Langer, Ph.D., Principal Investigator — Harvard U
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Bertisch SM, Legedza AR, Phillips RS, Davis RB, Stason WB, Goldman RH, Kaptchuk TJ. The impact of psychological factors on placebo responses in a randomized controlled trial comparing sham device to dummy pill. J Eval Clin Pract. 2009 Feb;15(1):14-9. doi: 10.1111/j.1365-2753.2008.00942.x. PMID 19239577
- [Background] Dawes P, Hopkins R, Munro KJ. Placebo effects in hearing-aid trials are reliable. Int J Audiol. 2013 Jul;52(7):472-7. doi: 10.3109/14992027.2013.783718. Epub 2013 Apr 18. PMID 23594421
- [Background] Labus J, Breil J, Stutzer H, Michel O. Meta-analysis for the effect of medical therapy vs. placebo on recovery of idiopathic sudden hearing loss. Laryngoscope. 2010 Sep;120(9):1863-71. doi: 10.1002/lary.21011. PMID 20803741
- [Background] Brown, J. A., Fowler, S. L., Rasinski, H. M., Rose, J. P., & Geers, A. L. (2013). Choice as a moderator of placebo expectation effects: Additional support from two experiments. Basic and Applied Social Psychology, 35(5), 436-444.
- [Background] Holmes EA, Ghaderi A, Harmer CJ, Ramchandani PG, Cuijpers P, Morrison AP, Roiser JP, Bockting CLH, O'Connor RC, Shafran R, Moulds ML, Craske MG. The Lancet Psychiatry Commission on psychological treatments research in tomorrow's science. Lancet Psychiatry. 2018 Mar;5(3):237-286. doi: 10.1016/S2215-0366(17)30513-8. No abstract available. PMID 29482764